CLINICAL TRIAL: NCT06910917
Title: Yeni Tanı Almış Meme Kanseri Hastalarına Uygulanan Roy Adaptasyon Temelli Hemşirelik Müdahalelerinin Psikolojik Dayanıklılık ve Psikososyal Uyum Üzerine Etkisi
Brief Title: The Effect of Roy Adaptation Model-Based Nursing Interventions on Psychological Resilience and Psychosocial Adjustment in Newly Diagnosed Breast Cancer Patients: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aytuğ Türk (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Aytuğ Türk, Dr., Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSKU-SBF-AT-03
Record Dates: First submitted 2024-12-08; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Psychosocial Adaptation; Psychological Resilience
Keywords: Breast cancer; Psychosocial Adaptation; Roy Adaptation Model; Nursing interventions; Psychological Resilience
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: After the research groups were formed, a six-session interview program was created for the participants in the experimental group. Individual goals were established by evaluating the psychosocial adjustment areas (physiological, self-concept, role function, interdependence) related to the disease and the stressors that could disrupt this adjustment (focus, characteristics). Nursing interventions were then applied in line with these goals.
  During the sessions, nursing and psychiatric nursing interventions based on the Roy Adaptation Model were implemented to address the anxiety experienced by individuals and the negative situations caused by that anxiety (such as psychoeducation, relaxation, mindfulness, and effective coping). Subjective goals were set for participants regarding the adaptive or maladaptive behaviors, attitudes, and thought patterns caused by the disease, and appropriate nursing interventions were applied from the Nursing Interventions Classification (NIC) system.
  Consid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roy Adaptation Model-Based Nursing Interventions Group (Experimental): A six-session program based on the Roy Adaptation Model was implemented for the experimental group, focusing on psychosocial adaptation (physiological, self-concept, role function, interdependence). Standard nursing interventions from NIC were applied, including enhancing coping, self-esteem, body image, and functional abilities. Outcomes were evaluated using NOC, and interventions were adjusted accordingly.
  Interventions: Behavioral: Roy Adaptation-Based Nursing Interventions
- Control Group (without any intervention) (No Intervention): Description: The control group received standard nursing care without additional interventions based on the Roy Adaptation Model. Their outcomes were monitored for comparison with the experimental group.

INTERVENTIONS:
Behavioral: Roy Adaptation-Based Nursing Interventions — After the research groups were formed, a six-session interview program was created for the participants in the experimental group. Individual goals were set for the participants in the experimental group by combining the evaluations of the areas related to the psychosocial adaptation brought by the disease (physiological, self-concept, role function, interdependence) and the stimuli that would disrupt the adaptation (focus, affecting and possible) and nursing interventions were determined in line with these goals.
  applied. In the sessions, nursing and psychiatric nursing interventions (psychoeducation, relaxation, awareness, effective coping) based on the Roy Adaptation Model were carried out for the negative situations caused by anxiety and anxiety experienced by individuals. It was applied to the participants as standard.
  Arms: Roy Adaptation Model-Based Nursing Interventions Group

SUMMARY:
Today, cancer has become a multifaceted problem whose diagnosis and treatment should be handled multidisciplinarily. In addition to being a medical-physical disease, cancer is a chronic phenomenon that involves many mental and psychosocial problems. Cancer patients develop various and different emotional, psychological and behavioral reactions during diagnosis, treatment, relapse and palliative periods. For this reason, holistic treatment and care of cancer patients should include medical, psychiatric and psychosocial dimensions together. Oncology, CLP and psychiatry nurses, who are important members of the team, have important duties in this regard. Accordingly, the study will be conducted with female individuals who applied to Ege University Tulay Aktas Oncology Hospital Psychooncology unit and were diagnosed with breast cancer within 6 months. The quasi-experimental method with pre-test post-test control group was used as the research method. In this context, the patients who applied to the relevant unit will be divided into two groups as experimental and control groups by simple randomization according to the order of application. SPSS 22 package program will be used in the evaluation of the data; statistical significance will be examined at 0.05 significance level. After the research groups are formed, a six-session interview program will be created for the participants in the experimental group. In the sessions, the most appropriate interventions based on the Roy Adaptation Model and the Nursing Interventions Classification System (Nursing Interventions Classification), including psychoeducation, adaptation to change, relaxation exercises, awareness, effective coping, problem solving, will be carried out for the negative situations that the disease and the disease may cause. At the end of each session, the evaluation of the interventions will be made according to the Nursing Outcomes Classification System. Individuals in the control group will not receive any intervention. The sub-concepts such as adaptation, stimulus, and behavior, which are considered and evaluated together within the conceptual framework of the Roy Adaptation model, are considered to be a highly suitable model for increasing psychosocial adaptation and psychological resilience in women newly diagnosed with breast cancer. The study data will be collected using the Individual Identification Form, Psychosocial Adjustment to Illness - Self-Report Scale and Psychological Resilience Scale. In addition to these scales that provide quantitative data, it is aimed to keep a researcher's diary during the sessions conducted by the researcher and to provide supportive data both for the evaluation of the needs and adaptation levels of the participants during the application process and for the evaluation of the application.

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers among women in terms of incidence and mortality rates and continues to be a major public health problem that poses a threat to women's health. According to 2020 statistics, female breast cancer has overtaken lung cancer as the most commonly diagnosed cancer. With 19.3 million new cases and 10.0 million deaths in 2020, compared to 18.1 million cases and 9.6 million deaths in 2018, the global cancer burden is increasing.

With this rise in breast cancer incidence, patients are exposed to many treatment methods and their side effects, such as hormonal drugs, surgical interventions, radiotherapy and chemotherapy, which cause intense stress due to the development of new treatment methods needed. Depending on the stage of the disease and individual characteristics of patients with breast cancer, several of these treatments may be preferred at the same time. Patients are exposed to many systemic effects of these interventions and treatment toxicity. While the aim of these treatments is to prolong the life of the patients and enable them to live with better quality of life, the physical, psychological, social well-being and daily vital functions of the patients may be negatively affected due to the prolonged duration of the interventions and the occurrence of systemic toxic effects. In addition to its high incidence, breast cancer is a serious disease due to its physical, psychological and emotional effects on women. It is important to identify and meet the information needs of women in this situation. Meeting these needs can improve the quality of life of these women by increasing their adaptation to the disease, improving their coping skills, accelerating their return to daily life, and reducing their anxiety and depression.

This long treatment process in breast cancer treatment involves a chronic recovery process that includes physical deficiencies, psychological, occupational and sexual problems, with periods of recovery and exacerbation, creating short and long-term adaptation difficulties. In the literature, there are studies indicating that many of the symptoms seen after chemotherapy can be significantly reduced by counseling, education, care and coaching practices given to patients, and that this can be provided by nurses who are in constant communication with patients. The main goal of the supportive role of the nurse is to help patients understand, cope with and adapt to distressing situations. It is very important for nurses to provide holistic care to women diagnosed with breast cancer, to address all the problems experienced by the patient and to provide counseling for them. Psychiatric and psychosocial care and treatment in patients with medical illnesses are reported to improve patient care and quality, reduce mortality and morbidity, decrease hospitalization time and general costs, and contribute to improvement and well-being. Developing the ability to recognize behaviors that indicate the presence of psychosocial problems and to manage them effectively will not only contribute to the well-being of patients, but also increase the motivation of nurses to address and intervene in psychosocial problems.

One of the many methods used for holistic care is interventions using models in practice. The Roy Adaptation Model (RAM), which is one of the widely used models in nursing, sees the person as a bio-psychosocial being in constant interaction with a changing environment. The environment includes focal, contextual and residual stimuli. The focal stimulus is the person's confrontation with the internal and external environment. The individual immediately resists these internal and external stimuli. Nurses aim to manage the focal stimulus first and then the contextual stimuli. Contextual stimuli are other stimuli that contribute to the focal stimuli and affect the current situation. Residual stimuli are implicit factors that influence the current situation. These are beliefs, behaviors and personal experiences. In the Roy Adaptation Model, which argues that nurses make interventions that facilitate the individual's adaptation to the environment, four different areas of adaptation are defined. These areas are physiological domain, self-concept domain, role function domain and interdependence domain. In these four adaptation domains, the nurse aims to improve the patient's interaction with the environment, develop adaptive behaviors and adapt to non-adaptive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Being a female aged 18 or older
* Having a confirmed breast cancer diagnosis within 0-6 months through clinical imaging and pathological examination
* Not having undergone surgery since the diagnosis or not having surgery planned within the study period (approximately 2 months) to exclude the impact of nursing care during surgical procedures

Exclusion Criteria:

* Non-primary breast cancer
* Presence of metastasis
* Receiving psychosocial treatment or therapy support
* Inability to attend sessions regularly
* Use of psychiatric medication within the last three months
* Having a low level of compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study included only female participants, as it focused on women newly diagnosed with breast cancer.
Enrollment: 44 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Psychosocial Adjustment to Illness Self-Report Scale (PAIS-SR) | Baseline (pre-test) and 6 weeks after the intervention (post-test)
  After obtaining the necessary permissions, women who participated in the study between December 2022 and November 2023 were provided with detailed face-to-face explanations about the research, and their written informed consent was obtained. The volunteers completed the scale forms in the hospital's psycho-oncology unit during six sessions, each lasting approximately 25-30 minutes.

SECONDARY OUTCOMES:
Psychological Resilience Scale (PRS) | Baseline (pre-test) and 6 weeks after the intervention (post-test)
  After obtaining the necessary permissions, women who participated in the study between December 2022 and November 2023 were provided with detailed face-to-face explanations about the research, and their written informed consent was obtained. The volunteers completed the scale forms in the hospital's psycho-oncology unit during six sessions, each lasting approximately 25-30 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The IPD (Individual Participant Data) will be shared upon request by contacting the responsible researcher.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 31.12.2-24-31.02.2025
Access Criteria: Researchers specializing in women and individuals with cancer will have access.